CLINICAL TRIAL: NCT01965873
Title: Enteral Nutrition for Treatment of Acute Pancreatitis - a Prospective, Randomized Clinical Trial
Brief Title: Enteral Nutrition in Acute Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Rijeka (Other)
Responsible Party: Principal Investigator, Goran Poropat, Medical doctor, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 062-0000000-0211
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Acute Pancreatitis
Keywords: Pancreatitis, Acute necrotizing; Enteral nutrition; Fasting; Complications; Mortality
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing; Fasting | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral nutrition (Experimental): In the enteral nutrition group a nasojejunal feeding tube will be placed via esophagogastroduodenoscopy and the position confirmed radiographically. Nutritional support will be started within 24 hours of enrollment, supplying daily 105 kJ (25 kcal)/kg, and 1.5 g/kg of protein based on ideal body weight. An elemental product for enteral nutrition will be infused at a rate of 25 ml/h, and increased by 10 ml/h every 6 hours, until the target rate of 100 ml/h will be achieved within 24-48 hours.
  Interventions: Dietary Supplement: Enteral nutrition
- Nil-by-mouth treatment (No Intervention): The nil-by-mouth treatment consists intravenous fluid replacement according to assessed needs via peripheral veins. This will include crystalloid (0.9% saline and 5% glucose), and colloid (10% hydroxyethyl starch and 3.5% plasma expander - haemaccel) solutions.

INTERVENTIONS:
Dietary Supplement: Enteral nutrition — Same as arm description
  Arms: Enteral nutrition

SUMMARY:
The purpose of this prospective randomised clinical trial is to compare beneficial and harmful effects of the use enteral nutrition versus a nil-by-mouth and intravenous fluid replacement principle of treatment in patients with moderate to severe acute pancreatitis (AP).

The hypothesis:

* enteral nutrition is no significantly better compared with the nil-by-mouth principle regarding mortality, incidence of local and systemic complications, length of hospital stay, and intensity of the inflammatory response in patients with moderate to severe AP
* enteral nutrition has the same safety as nil-by-mouth principle in patients with moderate to severe AP

DETAILED DESCRIPTION:
Patients with first attack of AP irrespective of etiology will be enrolled in the study, if they are eligible according to the following criteria:

Inclusion criteria:

* onset of symptoms consistent with AP within 72 hours before admission to the hospital
* an 3-fold elevation of serum amylase or serum lipase over the upper limit of normal
* APACHE II score 6 or more
* a signed informed consent

Exclusion criteria:

* patients < 18 years of age
* pregnant and breastfeeding women

ELIGIBILITY:
Inclusion Criteria:

* onset of symptoms consistent with AP within 72 hours before admission to the hospital
* an 3-fold elevation of serum amylase or serum lipase over the upper limit of normal
* APACHE II score 6 or more
* a signed informed consent

Exclusion Criteria:

* patients < 18 years of age
* pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
SIRS (Systemic Inflammatory Response Syndrome) | 4 weeks

SECONDARY OUTCOMES:
All-cause mortality | 4 weeks
Organ failure (cardiovascular, respiratory, renal) | 4 weeks
Local complications (pancreatic necrosis, fluid collections, pseudocyst, abscess) | 4 weeks
Local septic complications | 4 weeks
Other infections | 4 weeks
Inflammatory response (CRP on the first and third day) | First and third day of admission
Length of hospital stay | 4 weeks
Adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Davor Štimac, MD, PhD, Principal Investigator — Department of Gastroenterology, University Hospital Rijeka

REFERENCES:
- [Derived] Stimac D, Poropat G, Hauser G, Licul V, Franjic N, Valkovic Zujic P, Milic S. Early nasojejunal tube feeding versus nil-by-mouth in acute pancreatitis: A randomized clinical trial. Pancreatology. 2016 Jul-Aug;16(4):523-8. doi: 10.1016/j.pan.2016.04.003. Epub 2016 Apr 13. PMID 27107634